CLINICAL TRIAL: NCT01747122
Title: A Randomised Trial of Peri-operative Nerve Block and Continuous Infusion of Local Anaesthetic Via Wound Catheter Versus Epidural in Patients Undergoing Open Liver Resection.
Brief Title: The Effects of Local Infiltration Versus Epidural Following Liver Resection 2
Acronym: LIVER 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/R/SU/01 - LIVER 2 Trial
Record Dates: First submitted 2012-11-28; First posted 2012-12-11 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Open Liver Resection
Keywords: epidurals; wound catheters; liver resection; liver surgery
MeSH Terms: interventions — Injections, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wound catheter (Experimental): Wound catheter
  Interventions: Device: Wound catheter
- Epidural (Active Comparator): Standard epidural, pre-operative insertion, to be run for 48 hours
  Interventions: Device: Epidural

INTERVENTIONS:
Device: Wound catheter — Wound catheter, placed at end of procedure, prior to closure. To be kept in for 48 hours.
  Other Names: On-Q Painbuster
  Arms: Wound catheter
Device: Epidural
  Arms: Epidural

SUMMARY:
The investigators plan to compare epidurals versus wound catheters for effects on pain relief and recovery following open liver surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open hepatic resection for benign or malignant conditions.

Exclusion Criteria:

* Patients with contraindication to either epidural or wound catheter techniques.
* Inability to give written, informed consent.
* Jaundice (Bilirubin > 100 μmol/L)
* Liver resection combined with secondary surgical procedure.
* Age < 18 years
* Pregnant women
* patients on long term opiates for chronic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Length of stay | Measurement made on day of discharge which is expected to be on average bewteen 5 and 10 days after surgery.
  Number of days (to nearest half day) patients stay in hospital.

SECONDARY OUTCOMES:
Pain Scores | Performed daily at 0900 hours. On the day of surgery pain scores will be performed at 2, 6 and 12 hours post surgery.
  Visual analogue scores of pain experienced.
Molecular response to surgery | Days 0, 1 and 3
  HMGB1, RAGE and cytokines
Central Venous Pressure | During liver transection
  Mean Central Venous Pressure during liver transection will be quantified and compared between groups.
Estimated Blood Loss | Intra-operative
Operative field asessment | During liver transection
Pringle time | Intra-operative

OTHER OUTCOMES:
Quality of Life (EQ-5D) | Pre-operative, 2 weeks post-operative, 4-6 weeks post-operative
Morphine consumption | Day of surgery and postoperative days 1-7
IV Fluid volume | Day of Surgery and postoperative days 1-7
Complications | day of surgery and post-operative days 1-30
Post-operative blood tests (FBC, U&E, LFTs, coag) | Post-operative days 1-7

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Hughes, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Lothian, United Kingdom

REFERENCES:
- [Background] Revie EJ, McKeown DW, Wilson JA, Garden OJ, Wigmore SJ. Randomized clinical trial of local infiltration plus patient-controlled opiate analgesia vs. epidural analgesia following liver resection surgery. HPB (Oxford). 2012 Sep;14(9):611-8. doi: 10.1111/j.1477-2574.2012.00490.x. Epub 2012 Jun 10. PMID 22882198
- [Derived] Hughes MJ, Harrison EM, Peel NJ, Stutchfield B, McNally S, Beattie C, Wigmore SJ. Randomized clinical trial of perioperative nerve block and continuous local anaesthetic infiltration via wound catheter versus epidural analgesia in open liver resection (LIVER 2 trial). Br J Surg. 2015 Dec;102(13):1619-28. doi: 10.1002/bjs.9949. Epub 2015 Oct 8. PMID 26447461